CLINICAL TRIAL: NCT04727125
Title: Evaluating the Effects of Kangaroo Care in the NICU
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Craig Garfield, Professor of Pediatrics and Medical Social Sciences, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2019-2539
Record Dates: First submitted 2021-01-13; First posted 2021-01-27 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Kangaroo Care; Premature Birth; Fathers
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva is collected from infants, mothers, and fathers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main hypothesis of this study is that Kangaroo Father Care (KFC) will positively impact acute physiologic and long-term behavioral outcomes in infants, fathers, and families.

DETAILED DESCRIPTION:
Screening:

Participants will be recruited from the NICU at Prentice Women's Hospital. A member of the study team will screen all NICU patients for inclusion and exclusion criteria by reviewing electronic medical records. A screening and enrollment log will be kept to track families who have been approached and agreed or declined to participate in the study. The screening and enrollment log will be kept on a secure REDCap server housed by Northwestern University. Only the study team will have access to this log.

Kangaroo Care (KC) Intervention:

After enrollment, families will be scheduled to participate in two sessions of KC over two sequential days. The goal will be to schedule the KC sessions for the same time of day (i.e. morning, afternoon, or evening). However, if this is not possible given the parents', the sessions will be scheduled for any time of day that participating parents are able to visit their infant in the NICU. Each session will include two hours of continuous KC, with one day focused on Kangaroo Mother Care (KMC) and the other on Kangaroo Father Care (KFC), in a randomized order. These sessions will include continuous skin-to-skin holding of the infant by the parent, per standard of care protocol.

Physiologic Recording:

1) Infant: Prior to the first scheduled KC session, two wearable, wireless biosensors will be placed on the infant to continuously capture physiology measures including electrocardiogram (ECG), heart rate (HR), oxygen saturation (SpO2), body temperature, respiratory rate, movement, systolic blood pressure (BP-S), and others for the duration of the study. One device will be placed on the infant's chest or back. A second device will be placed peripherally, on the infant's leg, foot, arm, or hand. The devices are encapsulated in a medical-grade silicone and will be adhered to the infant's skin using a medical-grade adhesive, similar to the adhesives standardly used in the NICU. The biosensors will be left in place for up to 48 hours, but will be checked by study staff at least once every 24 hours to ensure skin integrity and signal quality. The adhesives will be changed between uses. 2) Parent: The same type of wearable, wireless biosensor will also be used to record 4 hours of continuous physiology including ECG, HR, temperature, movement, SpO2, and others in the infant's parents. The biosensor will be placed on the parent's chest 1 hour before the start of a scheduled KC session and worn for 1 hour preceding the scheduled KC session, during the 2-hour KC session, and for 1 hour after the completion of the KC session. The biosensor will be worn by the parents for approximately 4 hours in total.

Skin Monitoring:

Before and after the wearable biosensors are placed on the infant, the infant's skin integrity will be evaluated using the age-appropriate, NICU standard of care protocol for monitoring skin integrity. Study staff will take photographs of the skin at the site of biosensor placement before the biosensors are placed and after the biosensors are removed. Skin changes occurring while the biosensor is adhered to the infant's skin will be documented photographically. No faces will be photographed. The study team will consult the bedside care team within 1 hour for any ≥2 changes in skin integrity (based on the age-appropriate skin integrity scale score).

Video Monitoring:

In some patients, video monitoring of patient position and movement will be utilized during the study. This is an optional, additional part of the study in which families can choose to participate or not participate. For participating patients/families, a video camera will be mounted in the patient room for the duration of the KC sessions.

Saliva Sample Collection:

Saliva will be collected from enrolled infants and parents non-invasively to evaluate the effects of KFC on established biomarkers of stress (cortisol and testosterone) and father-infant bonding (oxytocin). Before, during, and after each KC session, saliva will be collected from the participating parent, and their infant. A trained member of the study team will collect saliva from infants using oral swabs made from an inert polymer and appropriately sized for an infant mouth (approximately 5 mm). Oral swabs will be taken from the infant immediately prior to beginning a KC session (T1), 30 minutes into the KC session (T2), and 30minutespost-session (T3). Parents will self-collect saliva samples at the time points outlined above, using an adult-sized oral swab. At T2, the trained study team member will be able to help the parent collect the saliva sample, if necessary, while the parent continues to hold their infant. This approach to salivary sample collection and biomarker analysis is similar to that established by previous studies of kangaroo care and takes into consideration the30-minute delay before cortisol reactivity in saliva.

Saliva Questionnaires:

When saliva is collected from parents at time points T1, T2, and T3, parents will also be asked to complete a brief saliva questionnaire. These questionnaires will take approximately five minutes each to complete and will be completed on paper or directly in REDCap, depending upon the participant's preferences. At T2, a study team member will be able to help the parent complete the survey, if necessary, while the parent continues to hold their infant. Data provided on surveys completed on paper will be transferred to secure REDCap forms by study staff and destroyed within 24 hours. All questionnaire data will be stored long term on the secure REDCap server housed by Northwestern University.

Psychosocial Questionnaires:

This study will employ psychosocial measures to capture the short- and long-term impacts of KFC. Specifically, validated measures of parenting confidence, relationship quality, infant bonding, and father involvement will be assessed via a set of paper or REDCap surveys administered in the NICU (short term) at baseline and the day before discharge (T-1) , and at home (long term) at 2 weeks (T+14) and 4 weeks (T+30) after discharge. Each of these sets of surveys will take approximately 30 minutes to complete. At baseline, each parent will complete the Revised Dyadic Adjustment Scale (RDAS) and the Postpartum Bonding Questionnaire (PBQ). At T-1, each parent will complete the RDAS , the PBQ, and the Parenting Sense of Competence Scale (PSOC). These questionnaires will be completed on paper or directly in REDCap, depending upon the participant's preferences. Data provided on surveys completed on paper will be transferred to secure REDCap forms by study staff and destroyed within 24 hours. At T+14 and T+30, each parent will complete the RDAS, the PBQ, the PSOC, and a Father Involvement Questionnaire. These questionnaires will be completed directly in REDCap only. Each parent will receive an email containing a link to their set of questionnaires at both post-discharge time points. All questionnaire data will be stored long term on the secure REDCap server housed by Northwestern University.

Wearable Sensor Data Collection:

The wearable sensor that will be used in this study can stream data continuously using near field communication (NFC) or Bluetooth technology. An encrypted laptop, iPad, or similar device will be left in the patient room and used to capture the continuous data stream from the wearable sensor. Additionally, wearable biosensors can include onboard memory, and physiologic streams may be recorded to this onboard memory until transfer to an encrypted laptop for analysis.

Standard of Care Data Collection:

In all patients in rooms where data from standard of care monitoring is recorded on the BedMaster system, this data will be used for comparison to data captured using the wearable sensors. In participants in rooms where this system is not available, the MediCollector system will be used to capture background data during the approximately 48-hour study.

ELIGIBILITY:
Inclusion Criteria:

* Infants: Infants who are born at Prentice Women's Hospital between 30 0/7 and 36 6/7 weeks gestation, are ≤20 days old at the time of enrollment, and do not meet any of the study's exclusion criteria will be eligible for participation in this study. Additionally, infants will only be included in this study if both of their biological parents are eligible and agree to participate.
* Parents: Parents who are ≥18 years of age, English speaking, expect mother and father to raise the infant together in the same household regardless of their marital status, and do not meet any of the study's exclusion criteria will be eligible for participation in this study. Additionally, family units will only be included in this study if both biological parents of the infant are eligible and agree to participate. Only English speaking parents will be included in this trial because the study questionnaires are only available in English.

Exclusion Criteria:

* Infants: Infants who are intubated or sedated, are receiving vasopressors or analgesics, have any congenital anomalies or skin abnormalities deemed likely to impact KC by clinical team, have received or are planned to receive surgical intervention, or are experiencing other symptoms or receiving other intervention that will impact the utilization of KC, wearable sensors, and/or oral swabs will be excluded from this study.
* Parents: Parents who are showing any signs of illness or taking corticosteroids or testosterone supplementation will be excluded from this study. Non-English speaking parents will also be excluded from this study because the questionnaires associated with this study are only available in English.

Ages: 1 Day to 20 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates (birth to less than 1 month) and adults (18 years and older)
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Infant Cardiorespiratory Stability | up to 48 hours, during scheduled skin-to-skin participation
  Heart rate (HR), oxygen saturation (SpO2), and HR variability (HRV) data collected before, during, and after KC will be combined to report infant cardiorespiratory stability.
Parent Physiologic Stress | up to 48 hours, during scheduled skin-to-skin participation
  Parent physiologic stress will be assessed through heart rate (HR) and HR variability (HRV) data collected before, during, and after KC.

SECONDARY OUTCOMES:
Accelerometry Accuracy | up to 48 hours, during scheduled skin-to-skin participation
  Accuracy of the biosensors to detect body position will be assessed through accelerometry data captured before, during, and after KC.
Infant Salivary Biomarker Analysis | Up to 4 hours. Before, during, and after each study skin-to-skin session
  Infant cortisol levels measured from saliva collected before, during, and after KC sessions will be used to assess infant stress response to KC.
Parent Stress Response | Up to 4 hours. Before, during, and after each study skin-to-skin session
  Paternal cortisol levels measured from saliva collected before, during, and after KC sessions will be used to assess parent stress response to KC.
Paternal Bonding | Up to 4 hours. Before, during, and after each study skin-to-skin session
  Paternal testosterone and oxytocin levels, measured in saliva collected before, during, and after KC, will be combined to report paternal bonding.
Parent Sense of Competency | An average of 4 weeks. Day before discharge, 2 weeks post discharge, 4 weeks post discharge
  Parents sense of competency will be assessed through parent scores on the Parenting Sense of Competence Scale (PSOC) administered longitudinally throughout study participation. The PSOC has 17 items and is scored on a 6 point Likert scale with a max of 102 and a min of 17, higher scores signal higher sense of parenting competency.
Parent Relationship Quality | An average of 6 weeks. Day of study consent, day before discharge, 2 weeks post discharge, 4 weeks post discharge
  Parents relationship satisfaction will be assessed through parent scores on the Revised Dyadic Adjustment Scale (RDAS) administered longitudinally throughout study participation. The RDAS is 14 items on a 5 or 6 point Likert scale, scores can range from 0-69 and a higher score signals greater relationship satisfaction.
Parent Bonding | An average of 6 weeks. Day of study consent, day before discharge, 2 weeks post discharge, 4 weeks post discharge
  Parent-infant bonding will be assessed through parent scores on the Postpartum Bonding Questionnaire (PBQ), administered longitudinally throughout study participation. The PBQ has 25 items scored on a 6 point Likert Scale with scores ranging from 0-125 and a lower score signaling better parent-infant bonding

CONTACTS AND LOCATIONS:
Overall Officials: Craig F Garfield, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern Medicine Prentice Women's Hospital, Chicago, Illinois

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT04727125/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT04727125/ICF_000.pdf